CLINICAL TRIAL: NCT06452654
Title: Anti-viral Action Against Type 1 Diabetes Autoimmunity
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Helmholtz Zentrum München (Industry); University Hospital Carl Gustav Carus (Other); Kinderkrankenhaus auf der Bult (Other); Skane University Hospital (Other); Universitaire Ziekenhuizen KU Leuven (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GPPAD-05-AVAnT1A
Record Dates: First submitted 2024-05-22; First posted 2024-06-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; T1D; Diabetes mellitus; Autoantigen; Prevention; at risk for developing type 1 diabetes; Juvenile diabetes; Autoimmune diabetes; Corona; COVID-19; Viral infection; Viral infection surveillance; Immune response; Metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; COVID-19; Virus Diseases | interventions — BNT162 Vaccine; Sodium Chloride; Solutions; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum (Active Comparator): Comirnaty® 3 µg Omicron XBB.1.5 or future new variant developments replacing current Comirnaty vaccines for children
  Suspension for injection, for intramuscular use
  1. st dose at age 6.0 to 7.0 months
  2. nd dose at least 3 weeks through to 6 weeks after 1st dose
  3. rd dose at least 8 weeks after 2nd dose (around age 8.5 to 11 months)
  Dose adjustment in case of COVID-19 infection.
  Interventions: Drug: Comirnaty Injectable Product
- Placebo (Placebo Comparator): 0.9 % Sodium Chloride Solution (saline) for intramuscular injection Dosing: three doses
  1. st dose at age 6.0 to 7.0 months
  2. nd dose at least 3 weeks through to 6 weeks after 1st dose
  3. rd dose at least 8 weeks after 2nd dose (around age 8.5 to 11 months)
  Interventions: Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: Comirnaty Injectable Product — Vaccination
  Other Names: Comirnaty 3µg/dose for children for 6 month - 4 years
  Arms: Verum
Drug: Sodium Chloride 0.9% Inj — Vaccination
  Other Names: Solution for Injection
  Arms: Placebo

SUMMARY:
The study GPPAD-05 AVAnT1A is a phase 4 clinical trial intending to enroll 2252 children, who will be randomly assigned to receive COVID-19 vaccination (Comirnaty® 3 μg Omicron XBB.1.5 or new variant Comirnaty vaccines ) or placebo from age 6 months.

The study is an investigator initiated, randomized, controlled, multicentre, multinational, primary prevention trial for children at increased risk of type 1 diabetes.

The primary objective is to determine whether vaccination of children with elevated genetic risk for type 1 diabetes against COVID-19 from 6 months of age reduces the cumulative incidence of islet autoantibodies or type 1 diabetes in childhood.

Secondary objectives are:

1. to determine whether vaccination against COVID-19 similarly reduces the cumulative incidence of multiple islet autoantibodies in childhood.
2. to determine whether vaccination against COVID-19 similarly reduces the cumulative incidence of type 1 diabetes in childhood and
3. to determine whether vaccination against COVID-19 similarly reduces the cumulative incidence of celiac disease-associated transglutaminase autoantibodies in childhood.

Further exploratory objectives are described in the study protocol.

Study participants will be identified through an ongoing study screening for genetic risk of type 1 diabetes using a polygenic risk score (NCT03316261).

Eligible participants will be enrolled at age 3.00 to 4.00 months (baseline visit).

Randomization to vaccine or placebo will occur at age 6.00 to 7.00 months at visit 2. Consent will be obtained by the custodial parents prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 3.00 and 4.00 months at the time of enrollment.
2. A high genetic risk (>10%) to develop islet autoantibodies by age 6 years as determined by a HLA DR/DQ genotype, polygenic risk score and first-degree family history of type 1 diabetes status.
3. Written informed consent signed by the custodial parent(s).

Exclusion Criteria:

1. Previous hypersensitivity to the excipients of the vaccine.
2. Any medical condition, concomitant disease or treatment that may interfere with the assessments or may jeopardize the participant's safe participation in the study. These include immune deficiencies, and conditions or treatments that lead to immune suppression.
3. Likely poor compliance due to expected change in residency.
4. Diagnosis of diabetes prior to recruitment or randomisation
5. Current use of any other investigational drug

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2252 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Persistent confirmed islet autoantibodies or type 1 diabetes | Through study completion, up to 6 years
  The primary outcome is the elapsed time from first vaccination to the development of persistent confirmed islet autoantibodies or type 1 diabetes.

SECONDARY OUTCOMES:
Persistent confirmed multiple islet autoantibodies | Through study completion, up to 6 years
  Elapsed time from first vaccination to persistent confirmed multiple islet autoantibodies;
Type 1 diabetes | Through study completion, up to 6 years
  Elapsed time from first vaccination to type 1 diabetes.
Persistent confirmed transglutaminase autoantibodies | Through study completion, up to 6 years
  Elapsed time from first vaccination to the development of persistent confirmed transglutaminase autoantibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Anette-G. Ziegler, Principal Investigator — Klinikum r.d.Isar of Technical University Munich and Institute for Diabetes Research, Helmholtz Munich, Heidemannstr.1, 80939 Munich, Germany
Locations (9):
- Medical University of Vienna, Dept. of Pediatric and Adolescent Medicine, Waehringer Gürtel 18-20, 1090 Vienna, Austria, Vienna, Austria
- University Hospitals Leuven, Faculty of Medicine, Catholic University of Leuven, Leuven, Belgium
- Germany (3):
  - Klinikum rechts der Isar of Technical University Munich and Institute for Diabetes Research, Helmholtz Munich, Munich, Bavaria
  - AUF DER BULT, Kinder- und Jugendkrankenhaus, Hanover, Lower Saxony
  - Klinik und Poliklinik f. Kinder und Jugendmedizin, Universitätsklinikum Carl Gustav Carus, Technische Universität Dresden, Dresden, Saxony
- Lund University Dep. of Clinical Sciences Malmo, Skane University Hospital SUS, Malmo, Sweden
- United Kingdom (3):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle